CLINICAL TRIAL: NCT03023982
Title: Ultrasound Guided PECs II (Pectoralis and Serratus Nerves) Block in Patients Undergoing a Thoracic Surgery
Brief Title: Pectoralis and Serratus Nerves Block in Thoracic Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Semionov Michael, Primary Investigator, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SOR 34516 CTIL
Record Dates: First submitted 2017-01-03; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia; Surgery; Block; Thoracic Injury
MeSH Terms: conditions — Bites and Stings; Thoracic Injuries | interventions — Bupivacaine; Ultrasonography; Thoracotomy; Analgesics, Opioid; Morphine; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pectoralic block group (Experimental): After general anesthesia, 40ml of 0.25% Bupivacaine Hydrochloride will be administered before procedure Thoracotomy. Block will be administrated between pectoralis minor and serratus anterior muscle at the 3rd and 4th rib., in assistance of ultrasound for visualization anesthetic injection point.
  Interventions: Drug: Bupivacaine Hydrochloride; Device: Ultrasound; Procedure: Thoracotomy; Drug: Opioids; Drug: NSAID
- Control group (Active Comparator): Patients in this group will receive standard pain control with opioids and NSAIDs
  Interventions: Procedure: Thoracotomy; Drug: Opioids; Drug: NSAID

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — 40 cc 0.25% of Bupivacaine Hydrochloride injection using ultrasound approach will be administered between pectoralis minor and serratus anterior muscle at the 3rd and 4th rib
  Other Names: Marcaine
  Arms: Pectoralic block group
Device: Ultrasound — All blocks will be done under ultrasound
  Other Names: Sonosite
  Arms: Pectoralic block group
Procedure: Thoracotomy — The patient population will include patients that undergo either open thoracotomy or thoracoscopy for anatomic and non-anatomic lung resection. The standard thoracoscopy approach in our institute includes three holes technic. There are two incisions of 1 cm and utility incision of 4 cm. The standard thoracotomy is posterior- lateral thoracotomy which divided the latissimus dorsi muscle but spears the serratus anterior muscle.
Drug: Opioids — standard pain control with opioids
  Other Names: Morphine
Drug: NSAID — standard pain control with NSAIDs
  Other Names: Perfalgan

SUMMARY:
A new conceptual regional anesthesia the PECs II block (modified pectoral and serratus nerves block) has been described for pain control after thoracic surgery, one of the indications to perform this method is analgesia for surgeries or procedures involving lateral chest wall

DETAILED DESCRIPTION:
The PECs I block was found to be very effective after breast cancer surgery and sub-pectoral prosthesis for pain control management.

This block is provided by injection into another myofascial plane, this time between pectoralis minor and serratus anterior muscle at the level of 3rd and 4th rib.PECs II block is simple in performance with a high success rate and minimal incidence of complications, especially, if used ultrasound approach that gives a good understanding of anatomy of the lateral thoracic wall.

In present clinical trial we are going to compare PECs block for pain control with traditional pain management techniques based on IV opioids and NSAIDs treatment in patient undergoing thoracic surgery in early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing thoracic surgery, older ≥18 years
2. Patients who meet criteria of ASA I-II-III class.

Exclusion Criteria:

1. Patients who will be unconscious or mentally incompetent
2. Patients refusal to participate in the study
3. ASA -IV -V
4. Patient with coagulopathy
5. Hemodynamically unstable (systolic BP < 90, HR > 100)
6. Allergy to local anesthetic drugs or opioids
7. Pregnant patient
8. History of opioid abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2017-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Comparison Visual Analog Score between groups | First 24 hours from the surgery
  First VAS after admission in PACU

SECONDARY OUTCOMES:
Total NSAIDs dosage (mg) in the PACU and department | First 24 hours from the surgery
  While the patient is in PACU
Length of hospital stay | up to 21 days
  Measuring time of at discharge from hospital
Total morphine dosage (mg) in the PACU and department | First 24 hours from the surgery
  While the patient is in PACU

IPD SHARING:
Plan to Share IPD: Undecided
will be decided later